CLINICAL TRIAL: NCT06603688
Title: Study on the Efficacy and Safety of Berberine, Minocycline, Esomeprazole, and Colloidal Bismuth Quadruple Therapy in the Initial Treatment of Helicobacter Pylori.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20232384-C-1
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection; Chronic Gastritis
Keywords: Berberine; Bismuth; Helicobacter Pylori; Minocycline
MeSH Terms: conditions — cyclopia sequence | interventions — Esomeprazole; Bismuth; Amoxicillin; Clarithromycin; Berberine; Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group：Minocycline+Berberine quadruple therapy (Experimental): 40mg of esomeprazole, 220mg of colloidal bismuth tartrate, 500mg of berberine hydrochloride, and 100mg of minocycline, taken orally twice daily for 14 days.
  Interventions: Drug: esomeprazole; Drug: Bismuth; Drug: Berberine; Drug: Minocycline
- control group：Amoxicillin+clarithromycin quadruple (Active Comparator): 40mg of esomeprazole, 220mg of bismuth tartrate colloid, 500mg of clarithromycin, and 1000mg of amoxicillin, taken orally twice a day for 14 days.
  Interventions: Drug: esomeprazole; Drug: Bismuth; Drug: Amoxicillin; Drug: clarithromycin

INTERVENTIONS:
Drug: esomeprazole — Esomeprazole 40mg, twice daily for 14 days.
Drug: Bismuth — Bismuth 220mg, twice daily for 14 days.
Drug: Amoxicillin — Amoxicillin 1000mg, twice daily for 14 days.
  Arms: control group：Amoxicillin+clarithromycin quadruple
Drug: clarithromycin — clarithromycin 500mg, twice daily for 14 days.
  Arms: control group：Amoxicillin+clarithromycin quadruple
Drug: Berberine — Berberine 500 mg, twice daily for 14 days
  Arms: experimental group：Minocycline+Berberine quadruple therapy
Drug: Minocycline — Minocycline 100 mg, twice daily for 14 days
  Arms: experimental group：Minocycline+Berberine quadruple therapy

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a quadruple therapy consisting of berberine hydrochloride, minocycline, esomeprazole, and colloidal bismuth tartrate for the first phase eradication of Helicobacter pylori. Assuming that the quadruple therapy of berberine hydrochloride, minocycline, esomeprazole, and colloidal bismuth tartrate is no less effective than the bismuth containing quadruple therapy of amoxicillin and clarithromycin. Patients diagnosed with Helicobacter pylori infection will be randomly assigned to one of the aforementioned treatments. During the 6-week follow-up, urea breath test, rapid urease test, or Helicobacter pylori fecal antigen test will be performed to confirm eradication.

The aim of this study is to evaluate the efficacy and safety of a quadruple therapy consisting of berberine hydrochloride, minocycline, esomeprazole, and colloidal bismuth tartrate for the first phase eradication of Helicobacter pylori. Assuming that the quadruple therapy of berberine hydrochloride, minocycline, esomeprazole, and colloidal bismuth tartrate is no less effective than the bismuth containing quadruple therapy of amoxicillin and clarithromycin. Patients diagnosed with Helicobacter pylori infection will be randomly assigned to one of the aforementioned treatments. During the 6-week follow-up, urea breath test, rapid urease test, or Helicobacter pylori fecal antigen test will be performed to confirm eradication.

DETAILED DESCRIPTION:
Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test，rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 13 and 17.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test，rapid urease test or helicobacter pylori stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection who did not receive Helicobacter pylori eradication treatment;
3. Patients are willing to receive eradication treatment.
4. Women of childbearing age were required to use medically acceptable contraceptive methods during and 30 days after the trial.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. Patients with contraindications or allergies to the study drug.
3. Severe organ damage and complications (such as liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases.
4. Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test),antibiotics or bismuth complexes (more than 3 times /1 month before screening).
5. Patients were diagnosed with gastroduodenal ulcer and MALTlymphoma.
6. Pregnant or lactating women.
7. Underwent upper gastrointestinal Surgery.
8. Patients with moderate to severe dysplasia or high degree of intraepithelial neoplasia.
9. Patients have symptom of dysphagia.
10. Evidence of bleeding or iron efficiency anemia.
11. A history of malignancy.
12. Drug or alcohol abuse history in the past 1 year.
13. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs,anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
14. Patients who has psychological problem or poor compliance.
15. Enrolled in other clinical trials in the past 3 months.
16. Refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
H pylori eradication rates | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative urea breath test，rapid urease test or helicobacter pylori stool antigen test 28 days after the end of treatment.

SECONDARY OUTCOMES:
symptoms effective rate | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment. Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%. Total score = frequency + severity. Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe

OTHER OUTCOMES:
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No